CLINICAL TRIAL: NCT03523780
Title: Is the Transfusion of Whole Blood Better for Resuscitation in Cesarean Delivery? A Retrospective Analysis of the Transfusion of Whole Blood Versus Component Therapy During Cesarean Delivery.
Brief Title: Transfusion of Whole Blood and Cesarean Delivery: A Retrospective Review
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 122016-079
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Obstetric Labor Complications
MeSH Terms: conditions — Obstetric Labor Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The rate of postpartum hemorrhage (PPH) has risen dramatically in the developed world, along with a rise in blood transfusion rates. The rate of cesarean delivery has increased dramatically in the past decade and is well over 30% in the United States. With an increase in primary and repeat cesarean delivery, comes the added risk of abnormal placentation, which can contribute to maternal and fetal morbidity and mortality via placenta accreta, increta, and percreta. The incidence of accreta has increased 10-fold over the past 50 years, becoming the most common reason for cesarean hysterectomy in highly industrialized countries. These conditions have tremendous impact on maternal outcomes.

Although whole blood (WB) contains all of the individual blood components, there are concerns for the use of WB due to the potential limitations such as the hemostatic efficacy of platelet after cold storage, the risk of hemolytic transfusion reaction following the transfusion of un-cross matched WB and the logistical issues in providing WB. Traditional obstetric transfusion protocols involve blood component therapy. Whole blood contains all components and could be more efficient for massive transfusion in obstetric hemorrhage. Trauma resuscitation protocols mimic whole blood in the 1:1:1 transfusion protocols of packed red blood cells to plasma to platelet ratio. It is difficult to compare trauma resuscitation to obstetric hemorrhage, but both can involve significant resuscitation and serious sequelae from unnecessary transfusion.

The use of WB instead of component therapy may reduce the multiple organ dysfunction rates due to the rapid resolution of shock and coagulopathy. Additionally, the number of donor exposure is important factor for the transfusion-related allergic reactions including severe systemic reactions such as anaphylaxis. Use of WB may decrease number of donor exposure. The secondary aim is to compare the incidence of 3 common adverse outcomes associated with the transfusion of blood products in subjects who receive whole blood versus component therapy.

Investigators hypothesize that the patients receiving WB will have fewer incidences of a) acute renal failure, b) acute heart failure and c) transfusion-related lung disease compared to those receiving component therapy.

DETAILED DESCRIPTION:
This is a retrospective cohort study. There is no research-related interventions. Data was collected retrospectively via the electronic medical records of the subjects who underwent cesarean delivery, and also received a blood transfusion during the intraoperative and postoperative periods between January 1, 2010 through December 1, 2016. Parkland Hospital Office of Research Administration pulled to data from eligible subjects' medical record based on ICD or CPT codes. Retrospective cohort was grouped as whole blood therapy and component therapy.

The data from the Electronic Medical Record pertaining to maternal characteristics includes demographic information, history of risk factors for PPH, prepartum and postoperative laboratory values, characteristic of cesarean section, type of the anesthesia utilized, Blood group, type and amounts of the blood products given, type of the components, how many overall units are given during the intraoperative period, need for an intraoperative hysterectomy, length of total hospital stay, evidences of hemolytic reaction caused by transfusion, the ICD 10 diagnosis of acute renal failure, acute heart failure due to volume overload, and transfusion-related lung disease (TRALI) on the discharge summary.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who underwent cesarean delivery
* Received a blood transfusion or blood component therapy

Exclusion Criteria:

* If sufficient information from the electronic record cannot be collected, those patients will be excluded.
* Subjects with pre-existing coagulation abnormalities such as hemophilia A, Von Willebrand's disease or any history of hereditary coagulopathies
* The utilization of the Massive Transfusion Protocol (MTP) intraoperatively
* Subjects with pre-existing renal failure, preexisting peripartum cardiomyopathy, or acute lung injury.
* Subjects who has transfusion of blood group O as non O recipient or received emergent uncross-matched blood in hospital admission or wrong blood transfusion.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female underwent cesarean delivery
Study Population: This is a retrospective study. Data retrospectively collected from medical record of the subjects underwent cesarean delivery and also received a blood transfusion or blood component therapy in the period between January 1, 2015 through January 1, 2016
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
Acute renal failure | During hospital stay approximately 2-3 week time frame
  Acute renal failure associated with the transfusion of blood products

SECONDARY OUTCOMES:
Acute heart failure | During hospital stay approximately 2-week time frame
  Acute heart failure associated with the transfusion of blood products
Transfusion-related lung disease | During hospital stay approximately 2-3 week time frame
  Transfusion-related lung disease following the transfusion of blood products

CONTACTS AND LOCATIONS:
Overall Officials: Seema Dave, MPH, Study Chair — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Hospital, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided